CLINICAL TRIAL: NCT06458322
Title: Prospective Changes in Quality of Life and Frailty in Chronic Kidney Disease Patients Transitioning to Home Versus In-Center Dialysis (QUALIFY CKD-to-HOME Study)
Brief Title: Quality of Life in Patients Transitioning to Home or In-Center Dialysis (QUALIFY CKD-to-HOME)
Status: Active, not recruiting | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: The Kidney Foundation of Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_2844
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Diseases; Quality of Life; Frailty; Dialysis; Home dialysis; In-center dialysis; Peritoneal dialysis; Home hemodialysis; Hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Home dialysis modality: Participants that determined peritoneal dialysis or home hemodialysis as their modality of treatment.
  Interventions: Other: Home dialysis or In-Center dialysis
- In-center dialysis modality: Participants that determined in-center hemodialysis as their modality of treatment.
  Interventions: Other: Home dialysis or In-Center dialysis

INTERVENTIONS:
Other: Home dialysis or In-Center dialysis — Initiation of dialysis with home dialysis (peritoneal dialysis or home hemodialysis) or in-center dialysis (hemodialysis)

SUMMARY:
The goal of this study is to evaluate quality of life (QoL) and frailty trajectories from advanced chronic kidney disease (CKD) to after dialysis initiation, specifically comparing patients choosing home dialysis and in-center hemodialysis.

The main questions it aims to answer are:

1. What is the trajectory of QoL in patients transitioning from advanced CKD to dialysis (up to 12 months after initiation) and how does these changes differ for patients oriented towards home dialysis and in-center hemodialysis?
2. Is the development of frailty after dialysis initiation less likely in patient pursuing home dialysis?
3. What is the variation in other PROMs and health outcomes (fatigue, anxiety & depression, general assessment, cognitive function) form advanced CKD to the first 12 months after dialysis initiation?
4. What are the predictors of severe decline in QoL, frailty and other important health outcomes (fatigue, cognition, anxiety & depression) during CKD G5 follow-up and after 12 months post dialysis initiation?

Participants will be ask to:

* Answer some questions and complete questionnaires each 3 months;
* Do a a grip test and a walking test each 6 months to evaluate their frailty;

DETAILED DESCRIPTION:
Background. Home dialysis is encouraged as the preferred therapy for people starting dialysis across Canada, with increased use of peritoneal dialysis (PD) and home hemodialysis (HHD) for patients with higher comorbidity burden. Dialysis modality selection is primarily a patient-centered choice. Modality selection should be mostly based on lifestyle and personal values. Despite the recognition of this patient-centered decision, most dialysis modality studies are based on mortality, hospitalization, and socioeconomic factors. There is a paucity of data to best inform patients of the expected changes in patient-reported outcomes measures (PROMs) such as quality of life (QoL), and the progression of their frailty status after dialysis initiation.

Objective. This study will fill this knowledge gap and evaluate QoL and frailty trajectories from advanced chronic kidney disease (CKD) to after dialysis initiation, specifically comparing patients choosing home dialysis and in-center hemodialysis (ICHD).

Design and Research Plan. Qualify CKD-to-Home is a prospective cohort study in 7 centers across Canada, with active patient-partner engagement. It is expected that around 200 patients will participate. Effort will be made to keep the ration of patients oriented towards home dialysis versus in-center at 1:2 or less.

Every 3 months participants will be followed, from estimated glomerular filtration rate (eGFR) <12 mL/min/1.73m2 and up to 12 months after dialysis start. They will be ask to complete questionnaires as the Kidney Disease Quality of Life (KDQOL-36), Quality of Life, the Hospital Anxiety and Depression Scale (HADS), the Standardized outcomes in Nephrology (SONG)-HD, Fatigue, the Medical Outcome Study- Social Support Survey (MOS-SSS), Social Support, the Montreal Cognitive assessment (MoCa), Cognitive Function, the Clinical Frailty Scale (CFS), the Fried Frailty Phenotype (FP) and the Gender-Related Variable for Health Research questionnaire (GVHR).

Analyse. Descriptive statistics will be used to report baseline characteristics for all patients. The KDQOL-36 components and domains, CFS, FI, HADS, SONG Fatigue instrument, feeling thermometer and MOCA, will be treated as continuous measures. Relationship between baseline scores will be assessed using Spearman correlation. Within patient changes in QoL, continuous frailty measures (CFS, FI), fatigue, depression & anxiety and general health will be described using generalized linear mixed effects models for repeated measures over time. Within patient changes in the proportion of patients classified as frail (vs. non-frail & pre-frail) using the FP with dichotomization will be analyzed in generalized linear mixed models with logistic links for binary repeated measures outcomes nested within centers. Missing data will be managed using multiple imputation by chained equations prior to proposed analyses.

Future directions. This study will help inform patients with advanced CKD on the trajectory of important patient-centered outcomes after dialysis initiation with different dialysis modality. Data from this study will be used to build on a mixed-methods approach with qualitative interviews of patients / caregiver to extend the reach of our understanding on PROMs (QoL) and frailty changes during the CKD to dialysis transition. Finally, the study results will guide stakeholders in the development of interventions that will mitigate risk of adverse outcomes for home dialysis patients at increased risk, as identified in our study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients followed in advanced CKD clinic;
* eGFR ≤12 mL/min/1.73m2 96;
* Understand English or French.

Exclusion Criteria:

* Orientation toward conservative treatment;
* Planned kidney transplantation < 6 months;
* Unable to provide consent due to severe cognitive or psychiatric disease;
* Previous treatment with dialysis > 3 month;
* Life expectancy < 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults followed in advanced chronic kidney disease clinics recruited from 7 centers across Canada
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Kidney Disease Quality of Life - 36 | From study inclusion until 12-months after dialysis start.
  Patients Scale from 0-100 (0 = poor, 100 = excellent).

SECONDARY OUTCOMES:
Change in Fried Frailty phenotype | From study inclusion until 12-months after dialysis start.
  5 components (slowness, weakness, weight loss, low physical activity, exhaustion) with classification as no-frail, pre-frail or frail.
Change in Clinical Frailty Scale | From study inclusion until 12-months after dialysis start
  Scale 1 (very fit) to 9 (terminally ill)
Change in Hospital Anxiety and Depression | From study inclusion until 12-months after dialysis start
  14 items scale (7 anxiety, 7 depression) with score >8 as cut-off for increased risk of depression and anxiety.
Change in Fatigue | From study inclusion until 12-months after dialysis start
  3 items questionnaire to assess fatigue and energy.
Change in Cognitive Function (MoCa) | From study inclusion until 12-months after dialysis start
  8 cognitive domains: attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations, and orientation with a possible score of 30 points.

CONTACTS AND LOCATIONS:
Overall Officials: Annie-Claire Nadeau-Fredette, MD, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada